CLINICAL TRIAL: NCT06579664
Title: Intermittent Theta Burst Stimulation on Cognitive Impairment of Cerebral Small Vessel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-A-2024044
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Small Vessel Diseases; Cognitive Impairment
Keywords: Cerebral Small Vessel Diseases; Cognitive Impairment; Intermittent Theta-Burst Stimulation; Personalized Brain Function Sector
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This trial was a randomized, single-center, double-blind, sham-controlled parallel trial. Participants were randomly assigned to receive iTBS stimulation or sham stimulation for 3 weeks in 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial is a double-blind design using simulants to ensure blinding. Participants will be randomly assigned to the iTBS and sham group according to the randomization codes that were generated by a computer program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iTBS group (Active Comparator)
  Interventions: Device: iTBS
- sham iTBS group (Sham Comparator)
  Interventions: Device: sham iTBS

INTERVENTIONS:
Device: iTBS — Participants in active group will receive iTBS stimulation in 50-Hz triplets at 5 Hz for 600 seconds per session (2 seconds on and 8 seconds off) at 90% of their resting motor threshold to the left dorsolateral prefrontal cortex (DLPFC).Each intervention day includes 4 sessions (1800 pulses/session) of stimulation delivering a total of 7200 active pulses. This treatment protocol will be conducted 15 consecutive days.
  Arms: iTBS group
Device: sham iTBS — Participants in the sham group will receive sham iTBS stimulation, which will use the same stimulation parameters, dosage, and duration as the active group, but will employ a sham coil. The sham coil is identical in appearance to the real stimulus coil and simulate the sound of a real stimulus, but do not produce a real stimulus.
  Arms: sham iTBS group

SUMMARY:
The cerebral small vessel diseases (CVSD) can cause severe and lasting damage to cognition function while the current available treatment of vascular cognitive impairment (VCI) is limited. The purpose of this study is to explore the feasibility, safety, and efficacy of intermittent Theta Burst Stimulation (iTBS) on cognitive impairment of cerebral small vessel disease.

DETAILED DESCRIPTION:
The cerebral small vessel diseases(CSVD) refers to any pathologic process that damages small end arteries, arterioles, venules, and brain capillaries. CVSD can cause severe and lasting damage to cognition function while the current available treatment of vascular cognitive impairment (VCI) is limited. Repetitive transcranial magnetic stimulation, a noninvasive neuromodulation treatment, has been proven effective for various neurological diseases such as depression, Parkinson's disease, poststroke movement disorders, and cognitive impairment. Theta-burst stimulation (TBS) has recently attracted broad attention as a form of accelerated repetitive transcranial magnetic stimulation that is more effective in achieving similar or higher therapeutic effects than conventional repetitive transcranial magnetic stimulation. The intermittent TBS (iTBS) has been considered to enhance cortical excitability. Personalized Brain Function Sector (pBFS) is a method that accurately delineate whole-brain personalized functional networks utilizing resting-state functional magnetic resonance imaging (MRI). The purpose of this study is to explore the efficacy and safety of iTBS under the guidance of pBFS in improving cognitive function in patients with CSVD.

This trial was a randomized, single-center, double-blind, sham-controlled parallel trial. The trial planned to enroll 58 patients with clinical evidence of CVSD and cognitive impairment, aged 45-85 years.

Participants were randomly assigned to receive iTBS stimulation or sham stimulation for 3 weeks in 1:1 ratio.

iTBS group: iTBS stimulation to the left dorsolateral prefrontal cortex (DLPFC), 1800 pulses /session, 4 sessions /day, as well as standard treatment and management according to the related guidelines.

sham iTBS group: mimicked iTBS stimulation at the same stimulation parameters, dose, and duration as the iTBS group with a sham coil, as well as standard treatment and management according to the related guidelines.

Follow up: Face to face interviews will be made on baseline, 15±7 days after randomization and 90±7 days after iTBS intervention.

The score of Montreal Cognitive Assessment Scale (MoCA) 90 days after iTBS intervention will be tested by the t-test or the Wilcoxon rank-sum test. The change of MoCA between baseline and 90 days after iTBS intervention will be tested by the two-sample t-test or the Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria：

1. Age 45-80 years old, with no limitation on sex.
2. Clinical evidence of CVSD as evidenced by one or more of:

   * White matter hyperintensity with Fazekas score ≥2
   * a lacunar stroke syndrome (e.g. pure motor stroke, pure sensory stroke, sensorimotor stroke, ataxic hemiparesis, or clumsy hand dysarthria syndrome) with a corresponding acute lacunar infarct on diffusion weighted imaging (DWl) for cases imaged (clinically) within 3 weeks of stroke or anatomically compatible lacunar infarct on fluid attenuated inversion recovery (FLAIR)/T1 MRI for cases imaged later after stroke (diameter≤1.5cm).
3. Independence of daily life (modified Rankin Scale score ≤2).
4. Mild vascular cognitive impairment (memory and/or other cognitive domain abnormalities lasting for at least 3 months) with a MoCA score of 10-22.
5. Routine, consistent medication for 4 weeks or more.

Exclusion Criteria:

1. History of stroke within previous 30 days, including cerebral infarction (diameter >15mm), cerebral hemorrhage, subarachnoid hemorrhage;
2. History of cerebral cortex infarction.
3. History of cerebrovascular malformation or aneurysmal subarachnoid hemorrhage, or discovery of an untreated aneurysm > 3mm.
4. Carotid or vertebral artery stenosis > 50% measured on North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria.
5. Possible amyloid cerebrovascular disease with at least 2 lobar hemorrhagic lesions (i.e., intracranial hemorrhage, cerebral microbleeds (CMB), cortical superficial siderosis, or convexal subarachnoid hemorrhage) measured on Boston Criteria 2.0; Or at least one lobar hemorrhagic lesion and at least one white matter feature (severe enlarged perivascular space in the centrum semiovale or multiple punctate white matter hyperintensities) without deep hemorrhagic lesion (cerebral hemorrhage or CMB) on T2* weighted MRI.
6. Recorded diagnosis of neurodegenerative diseases (e.g. Alzheimer's disease and Parkinson's disease).
7. Definite non-vasogenic white matter lesions (e.g. multiple sclerosis, cortical dysplasia in adults, metabolic encephalopathy).
8. Other psychiatric disorders diagnosed measured on the Diagnostic and Statistical Manual of Mental Disorders - V (DSM-V) diagnostic criteria; Or apparent suicidal intent.
9. Unable to tolerate MRI or contraindication to MRI (e.g., claustrophobia).
10. T1 or T2 weighted MRI shows focal brain injury.
11. Patients or first-degree relatives with a history of seizures.
12. Implanted pacemakers, vagus nerve stimulators, deep brain stimulators, or other metal medical devices.
13. Received transcranial magnetic stimulation therapy within previous 3 months.
14. Severe organic diseases with expected survival time <5 years, such as malignant tumor.
15. Women of child bearing potential, pregnant or breastfeeding.
16. Individual who have difficulty communicating verbally to the extent that they are unable to communicate, understand or follow instructions normally, and are unable to cooperate with treatment and evaluation.
17. Combined with alcohol and drug abuse history.
18. Unable to be cooperative and complete the follow-up due to geographical or other reasons.
19. Participated in other clinical trials.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montreal Cognitive Assessment Scale | at 90±7days after iTBS therapy
  Montreal Cognitive Assessment Scale (Beijing Edition) scores from 0 to 30. A higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Change from baseline in Mini-mental State Examination | at 90±7days after iTBS therapy
  Mini-mental State Examination (MMSE) scores from 0 to 30. A higher score indicates better cognitive function.
Change from baseline in verbal fluency test | at 90±7days after iTBS therapy
  Scoring of verbal fluency test (VFT) is based on the number of words produced by the participants from a category in a given time. A higher score indicates better cognitive function.
Change from baseline in trail making test | at 90±7days after iTBS therapy
  Scoring of color trial test (CTT) is based on time taken to complete the test and the number of wrong answers. Shorter the test time and less the mistakes, the better the outcome.
Change from baseline in Stroop Test | at 90±7days after iTBS therapy
  Scoring of Stroop Test is based on time taken to complete the test and the number of wrong answers. Shorter the test time and less the mistakes, the better the outcome.
Change from baseline in digital span test | at 90±7days after iTBS therapy
  Digital span test scores from 0 to 24. A higher score indicates better cognitive function.
Change from baseline in Hamilton Anxiety Scale | at 15±7days and 90±7days after iTBS therapy
  Hamilton Anxiety Scale (HAMA) scores from 0 to 56. A lower score indicates better emotional state.
Change from baseline in Hamilton Depression Scale | at 15±7days and 90±7days after iTBS therapy
  Hamilton Depression Scale (HAMD) scores from 0 to 68. A lower score indicates better emotional state.
Change from baseline in Pittsburgh sleep quality index | at 15±7days and 90±7days after iTBS therapy
  Pittsburgh sleep quality index (PSQI) scores from 0 to 21. A lower score indicates better sleep quality.
Change from baseline in The Short Physical Performance Battery(SPPB) | at 15±7days and 90±7days after iTBS therapy
  SPPB scores from 0 to 12. A higher score indicates better motor ability.
Change from baseline in The 5-level EuroQol five Dimensions Questionnaire | at 15±7days and 90±7days after iTBS therapy
  The 5-level EuroQol five Dimensions Questionnaire (EQ-5D-5L) scores from 0 to 25. A lower score indicates better life quality.
Change from baseline in 6 meter walk test | at 15±7days and 90±7days after iTBS therapy
  Scoring of 6 meter walk test is based on time taken to complete the test. A lower score indicates better motor ability.
Change from baseline in step-by-step walk test | at 15±7days and 90±7days after iTBS therapy
  Step-by-step walk test scores from 0 to 8. A lower score indicates better motor ability.
Change from baseline in 3-dimensional gait analysis (3D-IGA) | at 15±7days and 90±7days after iTBS therapy
  Gait features can be assessed with 3D-IGA providing rhythm, pace, phases, joint angle and other quantitative indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No